CLINICAL TRIAL: NCT05675787
Title: Medroxyprogesterone Acetate Plus Atorvastatin in Young Women With Atypical Endometrial Hyperplasia and Early Endometrial Carcinoma
Brief Title: Medroxyprogesterone Acetate Plus Atorvastatin in Young Women With Early Endometrial Carcinoma and Atypical Endometrial Hyperplasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Jianliu, Professor, Doctoral supervisor, Chief physician, Vice President, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022PHB416
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Atypical Endometrial Hyperplasia; Endometrial Carcinoma Stage I
Keywords: Endometrial Carcinoma; Atypical Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia; Endometrial Neoplasms | interventions — Medroxyprogesterone Acetate; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study: Control group and Experimental group;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): MPA + Atorvastatin
  Interventions: Drug: Medroxyprogesterone acetate + Atorvastatin
- Control groups (No Intervention): MPA

INTERVENTIONS:
Drug: Medroxyprogesterone acetate + Atorvastatin — MPA (at a dosage of 250-500 mg/day,) + Atorvastatin (at a dosage of 20 mg/day), by mouth,
  Arms: Experimental group

SUMMARY:
To explore the treatment efficacy of medroxyprogesterone acetate plus atorvastatin in patients with atypical endometrial hyperplasia (AEH) and early endometrial carcinoma (EEC) for conservative treatment.

DETAILED DESCRIPTION:
After diagnosed of AEH or EEC by hysteroscopy, patients meet the study criteria will be enrolled. The lipid content (lipid droplet, cholesterol and triglyceride) in endometrial lesion tissue was detected by Raman scattering instrument. And Age, height, weight, waistline, blood pressure, basic history of infertility and family cancer will be collected. Blood tests, including fasting blood glucose (FBG), fasting insulin (FINS), blood lipids, sex hormone levels, anti-müllerian hormone (AMH) and renal/liver function tests will be performed before treatment to evacuate their basic conditions. Each subject will receive body fat testing by Inbody 770.

Patients will receive MPA (Medroxyprogesterone acetate) 250-500 mg by mouth daily plus atorvastatin 20mg by mouth daily for at least 3 months. Then hysteroscopy will be used to evaluate the endometrial condition every 3 months, and intra-operative findings will be recorded. Complete response (CR) is defined as the reversion of endometrial atypical hyperplasia to proliferative or secretory endometrium; partial response (PR) is defined as regression to hyperplasia with or without atypic; stable disease (SD) is defined as the persistence of the disease; and progressive disease (PD) is defined as the appearance of higher pathological progression, or myometrial invasion, or extra-uterine metastasis. Continuous therapies will be needed in PR. Patients with PD will be recommended for hysterectomy.

For patients remained SD after 9 months of treatment but refused hysterectomy, a multiple disciplinary discussion would be held for individual case, and alternative treatment would be given. Three months of maintenance treatment will be recommended for patients with CR, and participants will be followed up for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed pathological diagnosis based upon hysteroscopy: histologically prove AEH or well-differentiated EEC G1 without myometrial invasion: 1. Untreated patients; 2. Patients with persistent lesions after one course (12 weeks) of progesterone therapy; 3. Patients who did not achieve complete remission after 2 courses (24 weeks) of progesterone therapy;
* No signs of suspicious extrauterine involvement on enhanced magnetic resonance imaging (MRI) or enhanced computed tomography (CT) or ultrasound
* Have a desire for remaining reproductive function or uterus
* Good compliance with adjunctive treatment and follow-up

Exclusion Criteria:

* Hypersensitivity or contradiction for using MPA or atorvastatin
* Pregnancy or potential pregnancy
* Confirmed diagnosis of any cancer in reproductive system
* Already diagnosed with hyperlipidemia and using lipid-lowering drugs
* Acute liver disease or liver tumor (benign or malignant) or renal dysfunction
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* With other factors of reproductive dysfunction;
* Strong request for uterine removal or other conservative treatment
* Smoker (>15 cigarettes a day)
* Drinker (>20 grams a day)

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathological cumulative complete response rate; | assessed up to 4 months
  3 to 4 months: From date of initial therapy until the date of CR or date of hysterectomy,

SECONDARY OUTCOMES:
Pathological cumulative complete response rate; | assessed up to 8 months
  From 6 to 8 months; From date of initial therapy until the date of CR or date of hysterectomy,
The lipid content (lipid droplet, cholesterol and triglyceride) in endometrial lesion tissue | assessed up to 4 months
  The lipid content (lipid droplet, cholesterol and triglyceride) in endometrial lesion
Overall complete response rate | up to 2 years
  Pathological response duration
Pathological response rate classified by different blood lipid level | up to 2 years;
  Pathological response rate classified by different blood lipid level
Relapse rate | up to 15 months after the end of treatment
  Relapse rate
Pregnancy rate | up to 15 months after the end of treatment
  Pregnancy rate
Toxic Side Effect | up to 3 months after the end of treatment
  Toxicity evaluation according to CTCAE 5.0 version.

CONTACTS AND LOCATIONS:
Locations (1):
- Wang Jianliu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No